CLINICAL TRIAL: NCT05006495
Title: Randomized Controlled Trial: Comparison of Radiological and Axial Pain Outcome Between C3-6 Open Door Laminoplasty and C3 Laminectomy With Cervical Laminoplasty
Brief Title: Comparison Between C3-6 Laminoplasty and C3 Laminectomy With Cervical Laminoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1610-136-804
Record Dates: First submitted 2021-07-30; First posted 2021-08-16 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Myelopathy Cervical; Kyphosis Post Surgical; Neck Pain; Ossification of Posterior Longitudinal Ligament; Cervical Spondylosis With Myelopathy
Keywords: Laminoplasty; Laminectomy
MeSH Terms: conditions — Neck Pain; Ossification of Posterior Longitudinal Ligament

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial, assigning subjects to two groups: C3 laminectomy with laminoplasty and C3-6 laminoplasty
Who Masked: Participant
Masking Description: Using a generator of www.randomization.com, 100 subjects randomized into blocks of 50 and 50. To reproduce this plan, use the seed 3169 along with the number of subjects per block/number of blocks and (case-sensitive) treatment labels as entered originally.
  and (case-sensitive) treatment labels as entered originally. After randomization of 100 subjects, additional 26 subjects randomized into blocks of 13 and13. To reproduce this plan, use the seed 5134 along with the number of subjects per block/number of blocks and (case-sensitive) treatment labels as entered originally.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C3 laminectomy with C4-6 laminoplasty (Experimental): Cervical myelopathy patients who underwent C3 laminectomy with laminoplasty.
  Interventions: Procedure: C3 laminectomy
- C3-6 laminoplasty (Active Comparator): Cervical myelopathy patients who underwent C3-6 laminoplasty.
  Interventions: Procedure: C3 laminoplasty

INTERVENTIONS:
Procedure: C3 laminectomy — C3 laminectomy preserving semispinalis cervicis inserted into the axis.
  Arms: C3 laminectomy with C4-6 laminoplasty
Procedure: C3 laminoplasty — Conventional C3-6 laminoplasty, resulting in injury of semispinalis cervicis.
  Arms: C3-6 laminoplasty

SUMMARY:
Investigators performed a prospective randomized controlled trial for comparing postoperative clinical and radiological outcomes between C3 laminectomy with laminoplasty and C3-6 laminoplasty.

DETAILED DESCRIPTION:
Cervical laminoplasty is widely performed surgical techniques to cervical myelopathy patients. But it is well known that C3-6 Cervical laminoplasty often results in injury of the semispinalis cervicis inserted into the axis, which possibly causes postoperative cervical kyphosis and neck pain. C3 laminectomy with cervical laminoplasty is the modified technique preserving the semispinalis cervicis to reduce such complications of conventional C3-6 laminoplasty.

There has been a number of retrospective studies comparing C3 laminectomy with laminoplasty and C3-6 laminoplasty, however, there's no prospective randomized controlled study yet. Investigators performed a prospective randomized controlled trial for comparing postoperative clinical and radiological outcomes between C3 laminectomy with laminoplasty and C3-6 laminoplasty. Primary end points include the C2-7 spine cobb anlge, Neck Disability Index(NDI) at postoperative 1~3 year

ELIGIBILITY:
Inclusion Criteria:

* Cervical stenosis patients with or without cervical myelopathy.

Exclusion Criteria:

* Metastatic cancer patients.
* Any combined fracture.
* Previous surgery to cervical spine.
* inflammatory joint disease
* psychiatric illness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen C, Li J, Liao Z, Gao Y, Shao Z, Yang C. C3 laminectomy combined with modified unilateral laminoplasty and in situ reconstruction of the midline structures maintained cervical sagittal balance: a retrospective matched-pair case-control study. Spine J. 2020 Sep;20(9):1403-1412. doi: 10.1016/j.spinee.2020.04.023. Epub 2020 May 6. PMID 32387294
- [Background] Kudo H, Takeuchi K, Wada K, Kumagai G, Tanaka S, Asari T, Araki R, Yokoyama T, Ishibashi Y. Ten-Year Long-term Results of Modified Cervical Double-door Laminoplasty With C3 Laminectomy Preserving the Semispinalis Cervicis Inserted Into the Axis Compared With Those of Conventional Cervical Laminoplasty. Clin Spine Surg. 2021 Apr 1;34(3):E147-E153. doi: 10.1097/BSD.0000000000001068. PMID 32941312
- [Background] Nakajima K, Nakamoto H, Kato S, Doi T, Matsubayashi Y, Taniguchi Y, Yoshida Y, Kawamura N, Nakarai H, Higashikawa A, Tozawa K, Takeshita Y, Fukushima M, Iizuka M, Ono T, Shirokoshi T, Azuma S, Tanaka S, Oshima Y. A Multicenter Observational Study on the Postoperative Outcomes of C3 Laminectomy in Cervical Double-door Laminoplasty. Clin Spine Surg. 2021 May 1;34(4):146-152. doi: 10.1097/BSD.0000000000001100. PMID 33086255
- [Background] Lee GW, Cho CW, Shin JH, Ahn MW. Which Technique Is Better Option for C3 Segment in Multilevel Open-Door Laminoplasty of the Cervical Spine?: Laminectomy Versus Laminoplasty. Spine (Phila Pa 1976). 2017 Jul 15;42(14):E833-E840. doi: 10.1097/BRS.0000000000001974. PMID 27851661
- [Background] Takeuchi K, Yokoyama T, Aburakawa S, Saito A, Numasawa T, Iwasaki T, Itabashi T, Okada A, Ito J, Ueyama K, Toh S. Axial symptoms after cervical laminoplasty with C3 laminectomy compared with conventional C3-C7 laminoplasty: a modified laminoplasty preserving the semispinalis cervicis inserted into axis. Spine (Phila Pa 1976). 2005 Nov 15;30(22):2544-9. doi: 10.1097/01.brs.0000186332.66490.ba. PMID 16284593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Started | 61 | 61
Completed | 51 | 58
Not Completed | 10 | 3

BASELINE CHARACTERISTICS:
Population: patients with more than postoperative 1year follow up were analysed.
Groups:
- Total: Total of all reporting groups
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty | Total
Number analyzed (Participants) | 51 | 58 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.4) | 58.3 (11.3) | 59.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 37 | 44 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease [Count of Participants; unit: Participants]
  Cerivcal spondylotic myelopathy | 30 | 31 | 61
  Ossification of posterior longitudinal ligament | 21 | 27 | 48
BMI [Mean (Standard Deviation); unit: Kg/m2] | 25.0 (3.0) | 25.5 (3.7) | 25.3 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: C2-C7 Lordosis
Description: Measuring C2-C7 lordosis angle by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: °
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
° | 11.0 (0.8) | 10.9 (0.8)

2. Primary Outcome: the Neck Disability Index (NDI)
Description: scores from 0 to 50 with 50 being the worst performance status related to neck pain.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
score | 12.8 (1.0) | 8.6 (1.0)

3. Secondary Outcome: C2-C3 Lordosis
Description: Measuring C2-C3 lordosis by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: °
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
° | 7.1 (0.5) | 3.2 (0.5)

4. Secondary Outcome: C4-C7 Lordosis
Description: Measuring C4-C7 lordosis by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: °
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
° | 3.9 (0.8) | 7.7 (0.7)

5. Secondary Outcome: Cervical Sagittal Vertical Axis (cSVA)
Description: Measuring cervical sagittal vertical axis by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
mm | 31.6 (1.4) | 25.5 (1.3)

6. Secondary Outcome: T1 Slope
Description: Measuring T1 slope by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: °
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
° | 25.8 (0.6) | 25.3 (0.6)

7. Secondary Outcome: T1 Slope Minus Cervical Lordosis
Description: Measuring T1 slope minus cervical lordosis by using standard lateral cervical x-ray series protocol with the patients standing in a neutral position and instructed to look straight ahead with knees locked.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: °
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
° | 15.0 (1.0) | 14.9 (0.9)

8. Secondary Outcome: C2-C3 Interlaminar Spontaneous Fusion
Description: Measuring the incidence of postoperative C2-C3 interlaminar spontaneous fusion by using standard lateral cervical x-ray series.
Time Frame: at 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
Participants | 5 | 26

9. Secondary Outcome: EuroQol Five-dimensional Questionnaire (EQ-5D) Scores
Description: Responses on a questionnaire with five dimensions, each comprised of five levels. Scores are revised into an index with a range from -0.59-1, with 1.00 indicating full health. The 243 possible health states on the EQ-5D are evaluated against a normal population using the time trade off method (TTO).
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
score | 0.661 (0.025) | 0.743 (0.024)

10. Secondary Outcome: Posterior Neck With Numering Rating Scale (NRS-N)
Description: Measuring pain intensity of the posterior neck with numeric rating scale (NRS), rated 1 to 10 with 10 being the most severe pain level.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
score | 2.8 (0.3) | 2.0 (0.3)

11. Secondary Outcome: Upper Limb Pain With Numering Rating Scale (NRS-L)
Description: Measuring pain intensity of the upper limb with numeric rating scale (NRS), rated 1 to 10 with 10 being the most severe pain level.
Time Frame: at 1, 2, 3 year (linear mixed-effect model analysis was used for repeated measurements)
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
score | 3.7 (0.4) | 2.8 (0.3)

12. Secondary Outcome: Estimated Intraoperative Blood Loss
Description: Measuring estimated intraoperative blood loss by using intraoperative records of anesthesiologists.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
cc | 169 (145) | 182 (159)

13. Secondary Outcome: Operative Time
Description: Measuring the time between start of the surgery (incision) and the finish of surgery (closure of the skin).
Time Frame: Intraoperative
Population: who completed 1-year to 3-year follow-up
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
Number analyzed (Participants) | 51 | 58
minutes | 126 (42) | 118 (40)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | C3 Laminectomy With C4-6 Laminoplasty | C3-6 Laminoplasty
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT05006495/Prot_SAP_000.pdf